CLINICAL TRIAL: NCT04007068
Title: FDG PET/CT Radiomics Analyses of Lung Cancer Patients Treated With Immunotherapy
Status: Completed | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: KME 117/02/17
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: RADIOMICS ANALYSIS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FDG PET/CT — FDG PET/CT baseline, month 1, month 4, month 10, than every 6 months

SUMMARY:
The investigators propose iRADIOMICS, a highly innovative and potentially clinical practice changing tool, which will allow for better management of patients undergoing immunotherapy. iRADIOMICS is based on in-depth interrogation of the molecular imaging (FDG PET/CT) data, extracting "invisible" information based on physical description of the imaging information. Based on the promising preliminary results of our pilot study, the investigators hypothesise that radiomics analyses of FDG PET/CT scans of patients treated with immunotherapy (iRADIOMICS) can better predict response to immunotherapy compared to the current standards (iRC). iRADIOMICS will be assessed in a prospective clinical study, involving 30 patients with metastatic non-small-cell lung cancer, treated with anti-programmed death-1 (anti-PD1) antibodies. Patients will undergo FDG PET/CT before the administration of anti-PD-1, at 1 month and 4 months after the administration. Afterwards, the patients will be imaged with FDG PET/CT every 6 months. Additionally, the patients will undergo diagnostic CT scan every 3 months to allow for comparison to the current standard (irRC).

DETAILED DESCRIPTION:
The investigators hypothesise that molecular imaging-based RADIOMICS analysis of FDG PET/CT data (termed iRADIOMICS) provides more information than standard anatomical imaging-based irRC analysis regarding the assessment of the effectiveness of immunotherapy and will have a stronger predictive power. It is widely accepted that molecular imaging (e.g. PET/CT) reflects changes in tissues much sooner than anatomical imaging (CT, MRI). Therefore, the investigators expect that an immunotherapy assessment tool based on FDG PET/CT should outperform anatomical-imaging-based irRC also timewise. Although the investigators do expect an initial increase in FDG PET uptake (mainly due to the metabolic activity of tumour infiltrating lymphocytes (TILs)), followed by a late decrease, the investigators argue that the predictive power of FDG PET can be even further increased by including an in-depth analysis of additional imaging features - the aforementioned "radiomics texture features". Many studies across different types of cancer have found a correlation between the presence of TILs and patient survival. Therefore the investigators expect that iRADIOMICS signature of responders will be different from the irRADIOMICS signature of non-responders to antiPD1 immunotherapy due to the different levels of TILs infiltration, different TILs spatial distribution within the tumour, and different composition of immunosuppressive tumour microenvironment containing different levels and spatial distribution of various immunosuppressive cells, such as myeloid-derived suppressive cells (MDSC), regulatory T cells (Treg), tumour-associated macrophages (TAM), regulatory dendritic cells (DCreg) and others 30. Thus the investigators anticipate that it might be possible to assess the response to immunotherapy at just one imaging time-point, preferably already in the pseudo-progression phase, thus much earlier than with irRC. Based on the assumption that irRADIOMICS might be able to detect differences in tumour immunosuppressive microenvironment, the investiagators further hypothesise that it might be also possible to predict, which patients are most likely to benefit from anti-PD1 immunotherapy already before the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Cytologically or histologically confirmed NSCLC with PD-L1 TPS ≥1% (confirmed by a validated test);
* Stage IVa, IVb or recurrent NSCLC (classification IASLC, 7th edition, 2009);
* Up to 10 metastases in multiple organ systems, or more than 10 metastases in more than two organ systems;
* No signs of active and/or untreated brain metastases;
* At least three measurable lesions;
* Progression after the first or second-line systemic therapy;
* WHO performance status 0-2 (ECOG criteria);
* Following the decision of multidisciplinary board that the patient is a candidate for treatment with pembrolizumab;
* FDG PET/CT performed up to 4 weeks prior to treatment;
* Performed diagnostic CT scans (thorax and abdomen) up to 4 weeks prior to treatment;
* Signed and dated written informed consent.

Exclusion Criteria:

Symptomatic and/or untreated brain metastases;

* History of other malignancies, except for the following: adequately treated basal or squamous cell carcinoma of the skin, curatively treated in situ carcinoma of the uterine cervix, other curatively treated solid tumour with no evidence of disease for ≥ 3 years;
* All contraindications for treatment with pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cytologically or histologically confirmed NSCLC patients with PD-L1 TPS ≥1% in stage IVa, IVb or recurrent NSCLC (classification IASLC, 7th edition, 2009) that are candidates for immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Correlation of iRADIOMICS with survival | 1.1.2017 - 31.12.2020
  To evaluate whether iRADIOMICS predicts response to immunotherapy better than irRC.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut of oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No